CLINICAL TRIAL: NCT00520806
Title: A Phase II/III, Multicenter, Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Relaxin in Subjects With Acute Heart Failure
Brief Title: Efficacy and Safety of Relaxin for the Treatment of Acute Heart Failure
Acronym: RELAX-AHF
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Corthera, Inc.(formerly BAS Medical, Inc.), a member of the Novartis group of companies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RLX.CHF.003
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-05

CONDITIONS: Heart Failure, Congestive
Keywords: Heart failure; Renal dysfunction; Relaxin; Vasodilator
MeSH Terms: conditions — Heart Failure; Renal Insufficiency | interventions — Relaxin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 48 hour iv infusion of placebo
  Interventions: Drug: Placebo
- Relaxin (Experimental): 48 hour iv infusion of relaxin at 30 ug/kg/day
  Interventions: Drug: Relaxin

INTERVENTIONS:
Drug: Relaxin — Intravenous infusion for 48 h at 30 ug/kg/day
  Arms: Relaxin
Drug: Placebo — Intravenous infusion for 48 h
  Arms: Placebo

SUMMARY:
Different doses of relaxin will be compared to placebo to determine efficacy and safety for the treatment of patients hospitalized with acute heart failure

DETAILED DESCRIPTION:
This is an international, randomized, double-blind, placebo-controlled, Phase II/III trial of intravenous recombinant relaxin for the treatment of signs and symptoms in patients hospitalized for acute decompensated heart failure. The Phase II pilot study has completed; the Phase III main portion of the trial is ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized for acute heart failure
* Dyspnea at rest or with minimal exertion
* Pulmonary congestion
* Able to provide informed consent
* Systolic blood pressure > 125 mmHg
* Impaired renal function defined as an eGFR of 30-75 mL/min/1.73m2

Exclusion Criteria:

* Use of other IV therapies for acute heart failure
* Fever or sepsis
* Recent major neurologic event
* Recent major surgery
* Recent acute coronary syndrome
* Other recent investigational drug use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1161 (Actual)
Dates: Start 2007-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Relief of dyspnea in acute heart failure | Up to day 5

SECONDARY OUTCOMES:
Days alive and out of hospital | Up to day 60
CV death or rehospitalization due to heart failure or renal failure | Up to day 60

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Severin, MD, Study Director — Novartis Pharmaceuticals
Locations (3):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Wayne State University/Detroit Receiving Hospital, Detroit, Michigan
- Heart Institute, Safed, Israel

REFERENCES:
- [Derived] Grand J, Miger K, Sajadieh A, Kober L, Torp-Pedersen C, Ertl G, Lopez-Sendon J, Pietro Maggioni A, Teerlink JR, Sato N, Gimpelewicz C, Metra M, Holbro T, Nielsen OW. Blood Pressure Drops During Hospitalization for Acute Heart Failure Treated With Serelaxin: A Patient-Level Analysis of 4 Randomized Controlled Trials. Circ Heart Fail. 2022 Apr;15(4):e009199. doi: 10.1161/CIRCHEARTFAILURE.121.009199. Epub 2022 Feb 21. PMID 35184572
- [Derived] Grand J, Miger K, Sajadieh A, Kober L, Torp-Pedersen C, Ertl G, Lopez-Sendon J, Pietro Maggioni A, Teerlink JR, Sato N, Gimpelewicz C, Metra M, Holbro T, Nielsen OW. Systolic Blood Pressure and Outcome in Patients Admitted With Acute Heart Failure: An Analysis of Individual Patient Data From 4 Randomized Clinical Trials. J Am Heart Assoc. 2021 Sep 21;10(18):e022288. doi: 10.1161/JAHA.121.022288. Epub 2021 Sep 13. PMID 34514815
- [Derived] Meyer S, Teerlink JR, Metra M, Ponikowski P, Cotter G, Davison BA, Felker GM, Filippatos G, Greenberg BH, Hua TA, Severin T, Qian M, Voors AA. Sex differences in early dyspnea relief between men and women hospitalized for acute heart failure: insights from the RELAX-AHF study. Clin Res Cardiol. 2017 Apr;106(4):280-292. doi: 10.1007/s00392-016-1051-4. Epub 2016 Nov 12. PMID 27838739
- [Derived] Felker GM, Teerlink JR, Butler J, Hernandez AF, Miller AB, Cotter G, Davison BA, Filippatos G, Greenberg BH, Ponikowski P, Voors AA, Hua TA, Severin TM, Unemori E, Metra M. Effect of serelaxin on mode of death in acute heart failure: results from the RELAX-AHF study. J Am Coll Cardiol. 2014 Oct 14;64(15):1591-8. doi: 10.1016/j.jacc.2014.05.071. PMID 25301463
- [Derived] Voors AA, Davison BA, Teerlink JR, Felker GM, Cotter G, Filippatos G, Greenberg BH, Pang PS, Levin B, Hua TA, Severin T, Ponikowski P, Metra M; RELAX-AHF Investigators. Diuretic response in patients with acute decompensated heart failure: characteristics and clinical outcome--an analysis from RELAX-AHF. Eur J Heart Fail. 2014 Nov;16(11):1230-40. doi: 10.1002/ejhf.170. Epub 2014 Oct 7. PMID 25287144
- [Derived] Teerlink JR, Cotter G, Davison BA, Felker GM, Filippatos G, Greenberg BH, Ponikowski P, Unemori E, Voors AA, Adams KF Jr, Dorobantu MI, Grinfeld LR, Jondeau G, Marmor A, Masip J, Pang PS, Werdan K, Teichman SL, Trapani A, Bush CA, Saini R, Schumacher C, Severin TM, Metra M; RELAXin in Acute Heart Failure (RELAX-AHF) Investigators. Serelaxin, recombinant human relaxin-2, for treatment of acute heart failure (RELAX-AHF): a randomised, placebo-controlled trial. Lancet. 2013 Jan 5;381(9860):29-39. doi: 10.1016/S0140-6736(12)61855-8. Epub 2012 Nov 7. PMID 23141816
- [Derived] Ponikowski P, Metra M, Teerlink JR, Unemori E, Felker GM, Voors AA, Filippatos G, Greenberg B, Teichman SL, Severin T, Mueller-Velten G, Cotter G, Davison BA. Design of the RELAXin in acute heart failure study. Am Heart J. 2012 Feb;163(2):149-55.e1. doi: 10.1016/j.ahj.2011.10.009. PMID 22305830
- [Derived] Voors AA, Davison BA, Felker GM, Ponikowski P, Unemori E, Cotter G, Teerlink JR, Greenberg BH, Filippatos G, Teichman SL, Metra M; Pre-RELAX-AHF study group. Early drop in systolic blood pressure and worsening renal function in acute heart failure: renal results of Pre-RELAX-AHF. Eur J Heart Fail. 2011 Sep;13(9):961-7. doi: 10.1093/eurjhf/hfr060. Epub 2011 May 28. PMID 21622980
- [Derived] Teerlink JR, Metra M, Felker GM, Ponikowski P, Voors AA, Weatherley BD, Marmor A, Katz A, Grzybowski J, Unemori E, Teichman SL, Cotter G. Relaxin for the treatment of patients with acute heart failure (Pre-RELAX-AHF): a multicentre, randomised, placebo-controlled, parallel-group, dose-finding phase IIb study. Lancet. 2009 Apr 25;373(9673):1429-39. doi: 10.1016/S0140-6736(09)60622-X. Epub 2009 Mar 28. PMID 19329178